CLINICAL TRIAL: NCT00002105
Title: Randomized, Comparative Trial of DOX-SL (Stealth Liposomal Doxorubicin Hydrochloride) Versus Bleomycin and Vincristine in the Treatment of AIDS-Related Kaposi's Sarcoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sequus Pharmaceuticals (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Model: Parallel | Purpose: Treatment
Other Study IDs: 134B; LTI-30-11
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1996-01

CONDITIONS: Sarcoma, Kaposi; HIV Infections
Keywords: Vincristine; Sarcoma, Kaposi; Liposomes; Doxorubicin; Drug Therapy, Combination; Acquired Immunodeficiency Syndrome; Bleomycin; Drug Carriers
MeSH Terms: conditions — Sarcoma, Kaposi; HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Doxorubicin; Liposomes; Bleomycin; Vincristine

INTERVENTIONS:
Drug: Doxorubicin hydrochloride (liposomal)
Drug: Bleomycin sulfate
Drug: Vincristine sulfate

SUMMARY:
To determine the efficacy of Stealth liposomal doxorubicin hydrochloride (DOX-SL) in the treatment of moderate to severe AIDS-related Kaposi's sarcoma (KS) by comparison with the established therapy BV (bleomycin/vincristine). To evaluate the safety and tolerance of DOX-SL compared to BV in a population of AIDS patients with moderate to severe KS.

DETAILED DESCRIPTION:
Patients are randomized to receive either DOX-SL or the BV combination. Infusions are given on day 1 and every 3 weeks for a total of six cycles. Kaposi's sarcoma lesions are evaluated prior to every cycle, at the end of the last treatment cycle, and 4 weeks following the end of the last treatment. Patients who respond to therapy will be followed every 2 months for up to 1 year. Patients must agree to have one or more representative KS lesions biopsied.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Prophylaxis for PCP, cryptococcal, and herpes infections, and antiretroviral therapy (e.g., AZT, ddC, ddI) provided these doses have been stable for at least 1 month.
* Maintenance therapy for tuberculosis, fungal, and herpes infections.
* Therapy for new episodes of tuberculosis, fungal, and herpes infection except with potentially myelotoxic chemotherapy.
* Foscarnet for cytomegalovirus infection.
* Erythropoietin.

Patients must have:

* Biopsy-proven, progressive, AIDS-related Kaposi's sarcoma, with any of the following:
* At least 15 mucocutaneous lesions.
* Six or more new lesions in the prior month.
* Documented visceral disease with at least five accessible cutaneous lesions.
* Documented anti-HIV antibody.
* No active opportunistic infection with mycobacteria, cytomegalovirus, toxoplasma, Pneumocystis carinii, or other microorganisms (if REQUIRING treatment with myelotoxic drugs).
* Life expectancy > 4 months.

NOTE:

* Patients who fail the BV combination or who relapse are eligible to enter the Liposome Technology open trial using DOX-SL alone.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Clinically significant cardiac disease.
* Confusion, disorientation, CNS symptoms, or peripheral neuropathy.

Concurrent Medication:

Excluded:

* Other cytotoxic chemotherapy.
* Colony-stimulating factors.
* Ganciclovir.

Patients with the following prior conditions are excluded:

* Prior neoplasms treated with extensive chemotherapy that, in the investigator's opinion, has led to irreversibly compromised bone marrow function.
* History of idiosyncratic or allergic reaction to anthracyclines, bleomycin, or vincristine.
* History of major psychiatric illness.

Prior Medication:

Excluded:

* Cytotoxic chemotherapy or interferon therapy within the past 4 weeks.
* More than one prior cycle of bleomycin/vincristine at any time.

Prior Treatment:

Excluded:

* Radiation or electron beam therapy within the past 3 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Beth Israel Hosp, Boston, Massachusetts
  - Mount Sinai Med Ctr, New York, New York
  - Twelve Oaks Hosp, Houston, Texas
  - Virginia Mason Research Center / Clinical Trial Unit, Seattle, Washington

REFERENCES:
- [Background] Stewart S, Jablonowski H, Goebel FD, L'Age M, Spittle M, Luthy R. Randomized comparative trial of DOXIL vs. Bleomycin and Vincristine in the treatment of AIDS-Related KS. Int Conf AIDS. 1996 Jul 7-12;11(Program Supplement):27 (abstract no LBB6026)